CLINICAL TRIAL: NCT04445441
Title: An Observational Study to Assess the Effectiveness of the Standard of Care (Hydroxychloroquine+Azythromicin or Chloroquine+Azythromicin) Recommended by the Ministry of Health for the Treatment of the Coronavirus Infection in Burkina Faso
Brief Title: An Observational Study to Assess the Protocol for the COVID-19 Treatment in Burkina Faso
Acronym: CHLORAZ
Status: Completed | Type: Observational
Sponsor: Centre Muraz (Other)
Responsible Party: Sponsor
Other Study IDs: IRSS-URCN-CM 001
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study to evaluate the effectiveness of the combinations Hydroxychloroquine + Azithromycin (HCQ-AZ) and Chloroquine + Azithromycin (CQ-AZ) in the treatment of Coronavirus (Covid-19) infection in Burkina Faso.

DETAILED DESCRIPTION:
All patients who received one of the two combinations will be included in the study and followed-up until the patient is discharged from the hospital. They will be seen daily during the period of their active clinical follow-up at the hospital. At each visit, the medical history since the last visit (including treatments taken), signs and symptoms in progress if any, will be collected. A nasopharyngeal swab will be collected on Day 0, 3, 7 and 14 and then on day 21 if he is still positive in order to assess the evolution of the viral load. However if until the end of the follow-up on D21 the test is still positive, the sampling will be continued until the patient become negative as recommended by the national standard of care for the Covid patients management in Burkina Faso.

In terms of safety, an ECG will be performed on day 0 prior to the treatment administration and this will be repeated on day 7 and day 14 and every week until it normalizes or the patient will be recommended to see a cardiologist to check the normalization of his ECG after discharge from hospital. Adverse events will be recorded including biological parameters (biochemistry and hematology) will be monitored, as well as changes in relevant laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 18 years treated according to the standard of care
* Willing to participate in the study by giving an informed consent

Exclusion Criteria:

* Patients under 18 years of age
* Not willing to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Any covid patient over 18 years treated according to standard of care
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Clearance of viral load | 14 days
  The impact of the treatment on virological clearance (viral load) post-treatment

SECONDARY OUTCOMES:
Safety of the treatment | 14 days
  This outcome will include the occurrence of adverse events including significant changes in the relevant biological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Halidou Tinto, PhD, Principal Investigator — IRSS - URCN
Locations (2):
- Burkina Faso (2):
  - Sourou Sanon University Hospital, Bobo-Dioulasso
  - Tingadogo University Hospital, Ouagadougou